CLINICAL TRIAL: NCT03655080
Title: Novel Approach of Pulsed Abraxane and Radiotherapy for Improving and Maintaining Ambulation After Cancer-Related Cord Compression
Brief Title: Pulsed Abraxane and Radiotherapy for Improving and Maintaining Ambulation After Cancer-Related Cord Compression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Pharmaceutical company decided to close study
Sponsor: Washington University School of Medicine (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201809175
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Results first posted 2021-10-18 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Cord Compression
MeSH Terms: conditions — Spinal Cord Compression | interventions — Radiotherapy; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- nab-Paclitaxel and Radiation Therapy (Experimental): * 10 fractions of 3Gy radiation therapy will be delivered.
  * A total of 4 chemoradiation blocks should be delivered ideally in consecutive days
  * On day 1 of the chemoradiation block, nab-paclitaxel is delivered in the morning followed by radiotherapy the latest possible and ideally at least 6 hours later (no earlier than 4 hours after the start of nab-paclitaxel)
  * On day 2, radiotherapy is delivered in the morning, ideally within 24 hours from the start of nab-Paclitaxel infusion the previous day
  * There will be 2 radiation fractions that won't be part of any chemoradiation block and can be placed anywhere before, after, or between blocks
  Interventions: Radiation: Radiation therapy; Drug: nab-Paclitaxel

INTERVENTIONS:
Radiation: Radiation therapy — Using the View Ray System
Drug: nab-Paclitaxel — * Dose 15 mg/m^2
  * Should be administered by IV over 30 minutes
  Other Names: Abraxane; Albumin-bound paclitaxel

SUMMARY:
The purpose of this research study is to look at a combination treatment of radiation therapy and a drug called Abraxane to treat epidural spinal cord compression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ≤ 37 points per the scoring system listed in the protocol
* Histologically or cytologically confirmed diagnosis of cancer not of CNS or spinal column origin.
* MRI or CT evidence of metastatic epidural spinal cord compression.
* Patients who have started 30 Gy in 10 fractions are not excluded as long as 4 doses of chemotherapy could potentially be given. This means the latest nab-paclitaxel can start is the morning of the third fraction of radiotherapy. Radiotherapy should ideally be delivered at least 6 hours after the nab-paclitaxel infusion started.
* At least 18 years of age.
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500 cells/mm3
  * Platelets ≥ 100,000 cells/mm3 (transfusion independent, defined as not receiving platelet transfusions within 7 days prior to blood draw)
  * Hemoglobin > 9.0 g/dL
  * Total bilirubin ≤ 1.5 mg/dL
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN
  * Alkaline phosphatase ≤ 2.5 x IULN (unless bone metastasis is present (< 5 x IULN) in the absence of liver metastasis)
  * Creatinine ≤ 1.5 mg/dL
* Women of childbearing potential (defined as a sexually mature woman who (1) has not undergone hysterectomy or bilateral oophorectomy or (2) has not been naturally postmenopausal for at least 24 consecutive months) must:

  * Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis) or agree to use, and be able to comply with, effective contraception without interruption, 28 days prior to starting treatment with nab-paclitaxel and while on study; and
  * Have a negative serum pregnancy test result at screening and agree to ongoing pregnancy testing during the course of the study and after the end of study therapy. This applies even if the subject practices true abstinence from heterosexual contact.
* Male subjects must practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions, and for 6 months following nab-paclitaxel discontinuation, even if he has undergone a successful vasectomy.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test prior to study entry.
* Known HIV-positivity on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with nab-paclitaxel. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Previous spinal cord radiotherapy that would overlap with the proposed treatment field.
* Spinal instability or bony retropulsion causing the cord compression. That is, mechanical, not tumor, cord compression. In these cases surgery may be indicated.
* Patients eligible for surgical decompression like laminectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiram A Gay, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nab-Paclitaxel and Radiation Therapy
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nab-Paclitaxel and Radiation Therapy
Number analyzed (Participants) | 2
Age, Continuous [Median (Full Range); unit: years] | 47.5 [37 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Ambulatory Status
Description: -Ambulatory status is categorized as paraplegic, not ambulatory, ambulatory with aid (for example, with assistive device like walker or crutches), and ambulatory without aid.
Time Frame: 1 month
Population: One participant was not evaluable for this outcome measure because the ambulatory status was not completed for the participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Paclitaxel and Radiation Therapy
Number analyzed (Participants) | 1
Participants
  Paraplegic | 0
  Not ambulatory | 1
  Ambulatory with aid | 0
  Ambulatory without aid | 0

2. Secondary Outcome: Ambulatory Status
Description: as for outcome 1
Time Frame: 3 months
Population: One participant was not evaluable for this outcome measure because the ambulatory status was not completed for the participant. One participant was not evaluable for this outcome measure because the participant died prior to the 3 month follow-up.
Arm/Group | Nab-Paclitaxel and Radiation Therapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Ambulatory Status
Description: as for outcome 1
Time Frame: 6 months
Population: Both participants expired prior to the 6 month follow-up.
Arm/Group | Nab-Paclitaxel and Radiation Therapy
Number analyzed (Participants) | 0

4. Secondary Outcome: Ambulatory Status
Description: as for outcome 1
Time Frame: 9 months
Population: Both participants expired prior to the 9 month follow-up.
Arm/Group | Nab-Paclitaxel and Radiation Therapy
Number analyzed (Participants) | 0

5. Secondary Outcome: Ambulatory Status
Description: as for outcome 1
Time Frame: 12 months
Population: Both participants expired prior to the 12 month follow-up.
Arm/Group | Nab-Paclitaxel and Radiation Therapy
Number analyzed (Participants) | 0

6. Secondary Outcome: Strength of Lower Extremities
Description: -Strength assessment is categorized as follows: 0/5=no contraction (worst); 1/5=muscle flicker, but no movement; 2/5=movement possible, but not against gravity (test the joint in its horizontal plane); 3/5=movement possible against gravity, but not against resistance by the examiner; 4/5=movement possible against some resistance by the examiner; 5/5=normal strength (best)
Time Frame: 1 month
Population: One participant was not evaluable for this outcome measure because the strength of lower extremities was not completed for the participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Paclitaxel and Radiation Therapy
Number analyzed (Participants) | 1
Participants
  0=no contraction | 0
  1=muscle flicker, but no movement | 0
  2=movement possible, but not against gravity (test the joint in its horizontal plane) | 0
  3=movement possible against gravity, but not against resistance by the examiner | 1
  4=movement possible against some resistance by the examiner | 0
  5=normal strength | 0

7. Secondary Outcome: Pain in the Irradiated Area" Measured on a Scale
Description: -Pain is measured on a scale between 0-10. 0=no pain (best) and 10=the greatest pain (worst)
Time Frame: 1 month
Population: One participant was not evaluable for this outcome measure because the pain scale was not completed for the participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Paclitaxel and Radiation Therapy
Number analyzed (Participants) | 1
Participants
  0 | 0
  1 | 0
  2 | 0
  3 | 0
  4 | 0
  5 | 1
  6 | 0
  7 | 0
  8 | 0
  9 | 0
  10 | 0

8. Secondary Outcome: Pain in the Irradiated Area Measured on a Scale
Description: -Pain is measured on a scale between 0-10. 0=no pain (best) and 10=the greatest pain (worst)
Time Frame: 3 months
Population: One participant was not evaluable for this outcome measure because the pain status was not completed for the participant. One participant was not evaluable for this outcome measure because the participant died prior to the 3 month follow-up.
Arm/Group | Nab-Paclitaxel and Radiation Therapy
Number analyzed (Participants) | 0

9. Secondary Outcome: Pain in the Irradiated Area Measured on a Scale
Description: -Pain is measured on a scale between 0-10. 0=no pain (best) and 10=the greatest pain (worst)
Time Frame: 6 months
Population: Both participants expired prior to the 6 month follow-up.
Arm/Group | Nab-Paclitaxel and Radiation Therapy
Number analyzed (Participants) | 0

10. Secondary Outcome: Pain in the Irradiated Area Measured on a Scale
Description: -Pain is measured on a scale between 0-10. 0=no pain (best) and 10=the greatest pain (worst)
Time Frame: 9 months
Population: Both participants expired prior to the 9 month follow-up.
Arm/Group | Nab-Paclitaxel and Radiation Therapy
Number analyzed (Participants) | 0

11. Secondary Outcome: Pain in the Irradiated Area Measured on a Scale
Description: -Pain is measured on a scale between 0-10. 0=no pain (best) and 10=the greatest pain (worst)
Time Frame: 12 months
Population: Both participants expired prior to the 12 month follow-up.
Arm/Group | Nab-Paclitaxel and Radiation Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From start of treatment through 28 days after completion of treatment (estimated to be 6 weeks) . Late toxicities for radiation therapy will be collected for 1 year after the end of radiation therapy (estimated to be 1 year and 2 weeks)
Arm/Group | Nab-Paclitaxel and Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 2/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-Paclitaxel and Radiation Therapy (N=2)
Paresthesia (Nervous system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-Paclitaxel and Radiation Therapy (N=2)
Blurred vision (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Fecal incontinence (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 2
Fatigue (General disorders) | 1
Thrush (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT03655080/Prot_SAP_000.pdf